CLINICAL TRIAL: NCT03320005
Title: EFFECTS OF RESISTANCE TRAINING ON THE PHYSICAL AND FUNCTIONAL RESPIRATORY PERFORMANCE OF ELDERLY
Brief Title: EFFECTS OF RESISTANCE TRAINING IN ELDERLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Daysi Tobelem (Other)
Responsible Party: Sponsor-Investigator, Daysi Tobelem, professor, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resist protocol
Record Dates: First submitted 2017-08-07; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Aging Disorder
Keywords: respiratory performance; quality of life; physical performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ResistanceTraining Group (Active Comparator): The RT program has the following features: 05 classes performing two weekly sessions; day shift; sessions with maximum duration of 1 (one) hour; 02 series; 08 to 12 repetitions; interval between sets of 01 to 02 minutes; exercises: bench press, seated leg press 45°, pull forward, Earth, rowing standing calf standing, power lifting, abdominal and development.
  Interventions: Other: Resistance training group
- Non training group (No Intervention): sedentary elderly

INTERVENTIONS:
Other: Resistance training group — Resistive exercises for legs and arms
  Arms: ResistanceTraining Group

SUMMARY:
This comes from a non-randomized clinical trial, which aims to check on elderly women the effects of a program of resistance training (TR) in physical performance, in respiratory functional capacity, on health and quality of life.

DETAILED DESCRIPTION:
Will be measured the strength of the respiratory muscles (Mip and Mep), peak expiratory flow (Peak-Flow), thoracic movements and abdominal movements, distance traveled in Incremental Shuttle Walk Test, grip strength manual, pulmonary leukocytes, biochemical parameters and indicators of quality of life and physical activity through the WHOQOL-old and IPAQ-short. The data will be tested against the distribution of the Gauss curve, by the shapiro-wilk test and, if they have a normal distribution (parametric) are expressed as mean and standard deviation, if not submit normal (non parametric) distribution will be expressed as median or range interquartílico. The first chance to compare the evolution of the group studied, will be applied to two-way ANOVA. If the distribution is abnormal, it will apply Mann-Whitney test. The multiple regression test will be used to compare the Mip and Mep with variables with the Peak-Flow, Thoracoabdominal mobility, distance traveled, immune competence, physical fitness and quality of life in the groups studied.

ELIGIBILITY:
Inclusion Criteria:

* 60 year old or more
* Do not have cardiac or respiratory diseases
* neurological, Musculoskeletal and other diseases preventing the practice of exercises
* not being a smoker; agree to participate in the study and signed an informed consent (IC); in the last six months preceding the evaluation did not have participated in physical activity program with the aim of improving physical performance.

Exclusion Criteria:

* Difficult to complete the tasks
* Acute diseases
* Refuse to continue the program

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Physical performance | Change from Baseline at 24 weeks
  distance traveled on ISWT

SECONDARY OUTCOMES:
quality of life | Change from Baseline at 24 weeks
  quality of life (WHOQOL-old)
respiratory muscle strength | Change from Baseline at 24 weeks
  respiratory pressures
Hand grip | Change from Baseline at 24 weeks
  Hand grip test

CONTACTS AND LOCATIONS:
Overall Officials: Dirceu Costa, PhD, Study Chair — Nove de Julho University

IPD SHARING:
Plan to Share IPD: No